CLINICAL TRIAL: NCT03548103
Title: Green Tea Extract for Obesity of Psychiatric Patients: a Double Blind Placebo-controlled Trial
Brief Title: Green Tea Extract for Obesity of Psychiatric Patients
Acronym: GEOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Lin, Shih-Ku, Chair, Department of Psychiatry, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10701-62-016
Record Dates: First submitted 2018-01-31; First posted 2018-06-07 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Tea

STUDY DESIGN:
Intervention Model Description: double blind placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green Tea Extract (Experimental): Green Tea Extract 500 mg per capsule
  Interventions: Dietary Supplement: Green tea extract
- Placebo (Placebo Comparator): Identical Placebo capsule
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Green tea extract — Green tea extract 500 mg tid for 16 weeks
  Arms: Green Tea Extract
Dietary Supplement: Placebo — Placebo tid for 16 weeks
  Arms: Placebo

SUMMARY:
Obesity or metabolic syndrome is becoming a global epidemic and common health problem, leading to the increase of associated comorbidities such as type 2 diabetes, cardiovascular disease, and certain cancers. This phenomenon is also a serious problem among psychiatric patients due to the increase use of second generation antipsychotics and mood stabilizers such as lithium or valproic acid. These metabolic abnormalities can be regarded as medical comorbidities, and have an impact not only on physical health and increased hospital length of stay, but also on a lower functional outcome, low self-esteem and poorer quality of life and non-compliance to antipsychotics. Green tea is one of the most popular beverages in the world and is believed to have beneficial effects in prevention and treatment of many diseases, such as cancer-prevention, adjunct to chemotherapy for malignancy, to reduce mental and physical stress and improve memory function, to increase bone mineral density, and to decrease body weight. Since weight gain is a common and undesirable side effect with psychiatric medications, the management of it becomes an important issue in clinical practice. In this clinical trial, we will use decaffeinated green tea extract to treat overweight patients with schizophrenia or bipolar disorder in a double-blind, placebo-controlled study design.

DETAILED DESCRIPTION:
Prevalence of obesity or metabolic syndrome and diabetes:

Obesity or metabolic syndrome is becoming a global epidemic and common health problem. The rising prevalence of obesity and associated comorbidities such as type 2 diabetes, cardiovascular disease, and certain cancers represents a major threat to public health worldwide. In a recent study in Asian populations, the result showed a strong association between BMI and prevalence of diabetes. From the results of a general population survey in Taiwan, the overall prevalence of obesity (body mass index (BMI) ≧ 27 kg/m2) in men and women was 19.2% and 13.4%, respectively, while the age-standardized prevalence of MS was 15.7% by the modified Adult Treatment Panel III criteria, 14.3% by the International Diabetes Federation for Chinese criteria and 16.4% by the metabolic syndrome criteria for Taiwanese. Their data also showed that the prevalence of obesity and metabolic syndrome significantly increased with age (trend test, p < 0.0001) in men and women. The risk of metabolic syndrome and its components increased significantly with BMI, and showed a marked increase with BMI≧24 kg/m2.

Prevalence of obesity or metabolic syndrome and diabetes in psychiatric patients:

The prevalence of MS among patients with schizophrenia or other psychotic disorder has been reported to be high, ranging from 24% to 43% in males and from 27% to 52% in females in previous large-scale investigations. These metabolic abnormalities can be regarded as medical comorbidities, and have an impact not only on physical health and increased hospital length of stay, but also on a lower functional outcome, low self-esteem and poorer quality of life and lead to non-compliant to antipsychotics.

In Taiwan, a large scale survey on 650 patients with schizophrenia or schizoaffective disorder from 36 community psychiatric rehabilitation centers or hospital-affiliated day hospitals in Taipei area revealed an overall metabolic syndrome prevalence of 34.9%, with 38.9% in female and 31.5% in male patients, respectively. The difference of metabolic syndrome prevalence between those patients and the general population was marked in male patients under 40 years of age and in female patients under 50. The authors suggested that BMI≧24 kg/m2 and age over 40 years old are two important risk factors of metabolic syndrome. Since the implementation of second generation antipsychotics (SGAs), especially clozapine, olanzapine or quetiapine, the metabolic syndrome prevalence exaggerated. Bai and her associates (2009) carried a large survey on 567 hospitalized of patients with schizophrenia under SGAs (clozapine =231, olanzapine n=94 and risperidone =242) for an average duration of 45.8+/-27.8 months, and revealed the prevalence of metabolic syndrome among all subjects was 23.8%. The clozapine group had a higher prevalence of metabolic syndrome (28.7%) than did the olanzapine (24.2%) and risperidone groups (19.5%) (P=0.039), and the clozapine group had lower levels of adiponectin (8.46+/-6.02 mg/mL) than did the olanzapine (10.26+/-4. 9 mg/mL) and risperidone groups (10.69+/-7.43 mg/mL) (P=0.001). The authors also found that adiponectin level was negatively correlated with BMI increase after initiation of SGAs treatment. Beside the increase use of SGAs, the use of mood stabilizers such as lithium or valproic acid in patients with bipolar disorder can also lead to body weight increment and metabolic syndrome.

Introduction of green tea:

Green tea is one of the most popular beverages in the world. It is made solely with the leaves of Camellia Sinensis that have undergone minimal oxidation during processing. Green tea is believed to have beneficial effects in prevention and treatment of many diseases, such as cancer-prevention and adjunct to chemotherapy for malignancy, to reduce mental and physical stress and improve memory function, to increase bone mineral density, and to decrease body weight. An epidemiological human study also showed that consumption of tea for more than 10 years led to a lower percentage of total body fat and smaller waist circumfluence. The anti-obesity effects of green tea are mainly attributed to its polyphenol content, in particular, epigallocatechin gallate (EGCG), which is most abundant in green tea and has been found to inhibit adipocyte proliferation and differentiation in in vitro studies.

Green Tea Extract studies in Taiwan:

In Taiwan, green tea extract (GTE) has been used to explore the effect on obese women by randomized, double-blind, placebo-controlled study design. Though the result showed that there was only a 0.3% reduction in body weight (0.15 kg) after 12 weeks of treatment with GTE in the study group, the GTE group had significant reduction in low-density lipoprotein (LDL)-cholesterol and triglyceride, and marked increase in the level of high-density lipoprotein (HDL)-cholesterol, adiponectin and ghrelin. In another study investigating insulin resistance type 2 diabetics patients, with no statistical difference was found in any measured variable between the decaffeinated GTE and placebo groups. However, there were some statistically significant within-group changes detected in items of reduction of waist circumference (WC), insulin resistance (HOMA-IR) index [fasting glucose (mmol/l) X fasting insulin (UI/l)/22.5], and insulin level, and a significant increase in the level of ghrelin. In an open label study, Tsai and his associates reported that more weight loss was found in the treatment group than the control (6.8 versus 2.3 kg; P <0.001) after 12-week use of green tea meal replacement formula product. Also, the treatment group had a greater changes in total cholesterol (185.2 versus 215.2 mg/dl; P=0.011) and low-density lipoprotein cholesterol (106.7 versus 127.6 mg/dl; P<0.005). Among completers only, the treatment group again lost more weight (6.8 kg; n=54 versus 0.8 kg; n=56; P =0.001) and had a greater reduced total body fat mass (7.6%; n=37 versus 0.5%; P=0.005). The authors concluded that green tea meal replacement formula contributes to the lower body weight and reduced low-density lipoprotein cholesterol level. Wu and his colleagues have carried out a cross-sectional survey of 1,210 epidemiologically sampled adults (569 men and 641 women) and found that habitual tea drinkers for more than 10 years showed a 19.6% reduction in body fat percentage (BF%) and a 2.1% reduction in waist-to-hip ratio (WPR) compared with non-habitual tea drinkers. The multiple stepwise regression models revealed that men, older age, higher BMI, and current smokers were positive factors for BF% and WHR. In contrast, longer duration of habitual tea consumption and higher total physical activity were negative factors for BF%. Longer duration of habitual tea consumption, higher socioeconomic status, and premenopausal status were negative factors for WHR.

Previous Study of GTE in Psychiatric patients:

Though there were a lot of researches regarding the use of GTE to treat metabolic syndrome or to decrease body weight across many countries, no one was focusing on the psychiatric patients. Katzman and his associates published a paper reporting 4 patients with resistant mood and anxiety disorder taking quetiapine and antidepressants, and used GTE by themselves for overweight and found that each patient had an unexpected decrease in total body fat mass, body fat percentage, and increase in lean body mass. Since weight gain is a common and undesirable side effect with psychiatric medications, especially the SGAs, the authors suggested the need for conducting controlled clinical trial using these agents to ameliorate these unwanted consequences.

In this clinical trial, the investigator will use decaffeinated green tea extract to treat overweight patients with schizophrenia or bipolar disorder in a double-blind, placebo-controlled study design.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with schizophrenia or mood disorders, followed at Taipei City Psychiatric Center will be the targeted study population. The subjects should fulfill the following criteria:

  1. Age between 20 to 65 years.
  2. Currently taking antipsychotics or mood stabilizers.
  3. BMI should be ≥ 27 kg/m2.
  4. Good adherence to medications as recorded by chart.
  5. Competent to understand the informed consent and have motivation to decrease their body weight.

Exclusion Criteria:

1. Unstable psychiatric symptoms or physical condition that may interfere the adherence of medication.
2. Medical conditions such as endocrine disease, heart disease, allergy or immunology disease, or impaired liver function (high aminotransferases, alanine, aspartate >80 IU/L or serum creatinine >2.5 mg/dl.
3. Pregnant or lactating women.
4. Childbirth within 6 months.
5. Management for weight control within 3 months.
6. Any other conditions deemed unsuitable for trial as evaluated by the physician-in-charge.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Body weight change in patients treated with psychotropic medications | 16 weeks
  Body weight decreas in kilogram after treatment

SECONDARY OUTCOMES:
Change of metabolic biochemistry profile composite | 16 weeks
  The change of Blood sugar in mg/dL, Triglyceride in mg/dL, Cholesterol in mg/dL, HDL-cholesterol in mg/dL, LDL-cholesterol in mg/dL, Hormone peptides Insulin in ng/mL, Leptin in ng/mL, Adiponectin in ng/mL and Ghrelin in ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City Hospital and Psychiatric Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No